CLINICAL TRIAL: NCT06003881
Title: An Open-Label, Expanded Access Program of Pozelimab in Patients With CD55-Deficient Protein-Losing Enteropathy (CHAPLE Disease)
Brief Title: Compassionate Use of Pozelimab in Patients With CD55-Deficient Protein-Losing Enteropathy
Acronym: CHAPLE Disease
Status: Approved for marketing | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: R3918-PLE-21110
Record Dates: First submitted 2023-08-14; First posted 2023-08-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: CD55-Deficient Protein-Losing Enteropathy

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Pozelimab — Subcutaneous (SC) administration
  Other Names: REGN3918

SUMMARY:
The program is to provide access to an experimental drug called pozelimab and to document the long-term safety of pozelimab in patients with Protein-Losing Enteropathy (PLE). CD55-deficient PLE/CHAPLE disease is a rare inherited disease of the immune system. This can be a life-threatening condition that is usually found when patients are children.

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical diagnosis of CD55-deficient PLE/CHAPLE disease (based on a history of PLE), confirmed by biallelic CD55 loss-of-function mutation detected by genotype analysis (frameshift, nonsense mutations) as defined in the protocol
2. Written informed consent from parent/guardian for minor patients
3. Written assent from minor patients as appropriate (eg, above the age of 6 years or the applicable age per local regulatory requirements)

Key Exclusion Criteria:

1. Patients who discontinued the prior pozelimab study due to safety or lack of efficacy
2. Considered by the treating physician as inappropriate for this program for any reason as defined in the protocol

NOTE: Other protocol defined inclusion / exclusion criteria apply

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult